CLINICAL TRIAL: NCT02179086
Title: Randomized Phase II Trial of Hypofractionated Dose-Escalated Photon IMRT or Proton Beam Therapy Versus Conventional Photon Irradiation With Concomitant and Adjuvant Temozolomide in Patients With Newly Diagnosed Glioblastoma
Brief Title: Dose-Escalated Photon IMRT or Proton Beam Radiation Therapy Versus Standard-Dose Radiation Therapy and Temozolomide in Treating Patients With Newly Diagnosed Glioblastoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: NRG Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NRG-BN001; NCI-2014-01072 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-BN001 (Other: NRG Oncology); NRG-BN001 (Other: CTEP); P50CA127001 (NIH); U10CA180868 (NIH); NCT02163135 (obsolete NCT alias)
Record Dates: First submitted 2014-06-27; First posted 2014-07-01 (Estimated); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Radiotherapy, Conformal; Radiotherapy, Intensity-Modulated; Photons; Radiation; Proton Therapy; Protons; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm A1 (control) (Active Comparator): Patients undergo standard-dose photon irradiation using 3D-CRT or IMRT QD, 5 days a week for 23 fractions plus a boost of 7 additional fractions.
  In all treatment arms, patients receive temozolomide PO QD on days 1-49 of radiation therapy. Beginning 4 weeks later, patients receive temozolomide PO QD on days 1-5. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: 3-Dimensional Conformal Radiation Therapy; Radiation: Intensity-Modulated Radiation Therapy; Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Drug: Temozolomide
- Arm A2 (control) (Active Comparator): Patients undergo standard-dose photon irradiation using 3D-CRT or IMRT as in Arm A1.
  In all treatment arms, patients receive temozolomide PO QD on days 1-49 of radiation therapy. Beginning 4 weeks later, patients receive temozolomide PO QD on days 1-5. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: 3-Dimensional Conformal Radiation Therapy; Radiation: Intensity-Modulated Radiation Therapy; Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Drug: Temozolomide
- Arm B (photon IMRT) (Experimental): Patients undergo dose-escalated and -intensified photon IMRT QD, 5 days a week for a total of 30 fractions.
  In all treatment arms, patients receive temozolomide PO QD on days 1-49 of radiation therapy. Beginning 4 weeks later, patients receive temozolomide PO QD on days 1-5. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: Intensity-Modulated Radiation Therapy; Other: Laboratory Biomarker Analysis; Radiation: Photon Beam Radiation Therapy; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Drug: Temozolomide
- Arm C (proton beam radiation therapy) (Experimental): Patients undergo dose-escalated and -intensified proton beam therapy QD, 5 days a week for a total of 30 fractions.
  In all treatment arms, patients receive temozolomide PO QD on days 1-49 of radiation therapy. Beginning 4 weeks later, patients receive temozolomide PO QD on days 1-5. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Radiation: Proton Beam Radiation Therapy; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Drug: Temozolomide

INTERVENTIONS:
Radiation: 3-Dimensional Conformal Radiation Therapy — Undergo standard-dose 3D-CRT
  Other Names: 3-dimensional radiation therapy; 3D Conformal; 3D CONFORMAL RADIATION THERAPY; 3D CRT; 3D radiotherapy; 3D-CRT; Conformal Therapy; Radiation Conformal Therapy; Radiation, 3D Conformal; Three dimensional external beam radiation therapy (procedure)
  Arms: Arm A1 (control); Arm A2 (control)
Radiation: Intensity-Modulated Radiation Therapy — Undergo standard-dose IMRT
  Other Names: IMRT; Intensity modulated radiation therapy (procedure); Intensity Modulated RT; Intensity-Modulated Radiotherapy; Radiation, Intensity-Modulated Radiotherapy
  Arms: Arm A1 (control); Arm A2 (control)
Radiation: Intensity-Modulated Radiation Therapy — Undergo dose-escalated and -intensified photon IMRT
  Other Names: IMRT; Intensity modulated radiation therapy (procedure); Intensity Modulated RT; Intensity-Modulated Radiotherapy; Radiation, Intensity-Modulated Radiotherapy
  Arms: Arm B (photon IMRT)
Other: Laboratory Biomarker Analysis — Correlative studies
Radiation: Photon Beam Radiation Therapy — Undergo dose-escalated and -intensified photon IMRT
  Other Names: External beam radiation therapy using photons (procedure); Photon; Photon EBRT; Photon External Beam Radiotherapy; PHOTON Therapy; Radiation, Photon Beam
  Arms: Arm B (photon IMRT)
Radiation: Proton Beam Radiation Therapy — Undergo dose-escalated and -intensified proton beam radiation therapy
  Other Names: External beam radiation therapy protons (procedure); External Beam Radiotherapy (protons); PBRT; Proton; Proton EBRT; Proton External Beam Radiotherapy; Proton Radiation Therapy; PROTON Therapy; Radiation, Proton Beam
  Arms: Arm C (proton beam radiation therapy)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Drug: Temozolomide — Given PO
  Other Names: CCRG-81045; Gliotem; Imidazo[5,1-d]-1,2,3,5-tetrazine-8-carboxamide, 3, 4-dihydro-3-methyl-4-oxo-; M & B 39831; M and B 39831; Methazolastone; RP-46161; SCH 52365; Temcad; Temizole; Temodal; Temodar; Temomedac; TMZ

SUMMARY:
This randomized phase II trial studies how well dose-escalated photon intensity-modulated radiation therapy (IMRT) or proton beam radiation therapy works compared with standard-dose radiation therapy when given with temozolomide in patients with newly diagnosed glioblastoma. Radiation therapy uses high-energy x-rays and other types of radiation to kill tumor cells and shrink tumors. Specialized radiation therapy that delivers a high dose of radiation directly to the tumor may kill more tumor cells and cause less damage to normal tissue. Drugs, such as temozolomide, may make tumor cells more sensitive to radiation therapy. It is not yet known whether dose-escalated photon IMRT or proton beam radiation therapy is more effective than standard-dose radiation therapy with temozolomide in treating glioblastoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine if dose-escalated and -intensified photon IMRT or proton beam therapy (using a dose-per-fraction escalation with simultaneous integrated boost) with concomitant and adjuvant temozolomide improves overall survival, as compared to standard-dose photon irradiation with concomitant and adjuvant temozolomide.

SECONDARY OBJECTIVES:

I. To indirectly compare dose-escalated and -intensified photon IMRT to dose-escalated and -intensified proton beam therapy in terms of overall survival.

II. To indirectly compare and record toxicities of dose-escalated and -intensified photon IMRT versus dose-escalated and -intensified proton beam therapy and directly compare the toxicities of these approaches versus standard-dose photon irradiation on the backbone of concomitant and adjuvant temozolomide.

III. To determine if dose-escalated and -intensified IMRT or proton beam therapy (using a dose-per-fraction escalation with simultaneous integrated boost) with concomitant and adjuvant temozolomide improves perceived cognitive symptom severity, as compared to standard-dose photon irradiation with concomitant and adjuvant temozolomide.

IV. To determine if dose-escalated and -intensified photon IMRT or proton beam therapy (using a dose-per-fraction escalation with simultaneous integrated boost) with concomitant and adjuvant temozolomide improves neurocognitive function, as compared to standard-dose photon irradiation with concomitant and adjuvant temozolomide.

V. To indirectly determine if dose-escalated and -intensified proton beam therapy with concomitant and adjuvant temozolomide improves perceived cognitive symptom severity, as compared to dose-escalated and -intensified photon IMRT, and to directly compare symptom burden with these approaches versus standard-dose photon irradiation on the backbone of concomitant and adjuvant temozolomide.

VI. To indirectly determine if dose-escalated and -intensified proton beam therapy with concomitant and adjuvant temozolomide improves neurocognitive function, as compared to dose-escalated and -intensified photon IMRT, and to directly compare neurocognitive function with these approaches versus standard-dose photon irradiation on the backbone of concomitant and adjuvant temozolomide.

EXPLORATORY OBJECTIVES:

I. Tissue banking for future translational science projects that will be determined based on the state of the science at the time the primary endpoint is reported and will be submitted to National Cancer Institute (NCI) for review and approval.

II. To prospectively compare CD4 lymphopenia between dose-escalated and intensified proton beam therapy, dose-escalated and -intensified photon IMRT, and standard-dose photon irradiation and determine whether CD4 lymphopenia impacts overall survival.

III. To explore the most appropriate and clinically relevant technological parameters to ensure quality and effectiveness throughout radiation therapy processes, including imaging, simulation, patient immobilization, target and critical structure definition, treatment planning, image guidance and delivery.

IIIa. To establish feasibility and clinical relevancy of quality assurance guidelines.

IIIb. To evaluate efficacy of quality assurance tools. IV. To explore the most appropriate and clinically relevant advanced and standard magnetic resonance imaging (MRI) imaging parameters.

IVa. To evaluate the feasibility of differentiating pseudo-progression and true progression in a multi institutional setting using magnetic resonance (MR) diffusion and perfusion imaging.

IVb. To evaluate for early, imaging biomarkers of response and overall survival.

OUTLINE: Patients are assigned to 1 of 2 groups depending on enrolling institution. Within each group, patients will be randomized 1:2 in favor of the experimental arms.

GROUP I (PHOTON IMRT CENTERS): Patients are randomized to 1 of 2 treatment arms.

ARM A1: Patients undergo standard-dose photon irradiation using 3-dimensional conformal radiation therapy (3D-CRT) or IMRT once daily (QD), 5 days a week for 23 fractions plus a boost of 7 additional fractions.

ARM B: Patients undergo dose-escalated and -intensified photon IMRT QD, 5 days a week for a total of 30 fractions.

GROUP II (PROTON CENTERS): Patients are randomized to 1 of 2 treatment arms.

ARM A2: Patients undergo standard-dose photon irradiation using 3D-CRT or IMRT as in Arm A1.

ARM C: Patients undergo dose-escalated and -intensified proton beam radiation therapy QD, 5 days a week for a total of 30 fractions.

In all treatment arms, patients receive temozolomide orally (PO) QD on days 1-49 of radiation therapy. Beginning 4 weeks later, patients receive temozolomide PO QD on days 1-5. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 1 year, every 4 months for 1 year, and then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* PRIOR TO STEP 1 REGISTRATION
* A diagnostic contrast-enhanced MRI (no other scan type allowed) of the brain must be performed postoperatively; the residual enhancing tumor and/or resection cavity must have a maximal diameter of 5 cm or less; the tumor diameter will be the greatest diameter as measured on the contrast-enhanced postoperative MRI and will include residual disease and/or the postoperative surgical cavity as appropriate

  * The postoperative brain MRI should be obtained within 72 hours of resection; if it is not obtained within 72 hours post-resection, then an MRI obtained 2 weeks or longer after surgery is required and can be utilized to ensure maximal diameter of residual tumor and/or resection cavity is 5 cm or less
  * For cases where a gross total resection of enhancing tumor is performed, but postoperative surgical cavity is NOT identifiable, the patient will be excluded from the trial
* Tumor tissue must be available for submission for central pathology review

  * Timing requirements:

    * If MGMT has been assessed locally by LabCorps or MD Anderson Cancer Center Molecular Diagnostics Lab (MDACC-MDL):

      * Tissue for central pathology review and central MGMT assessment and the official LabCorps or MDACC-MDL MGMT result must be received by the NRG Oncology Biospecimen Bank on or before postoperative calendar day 40
      * The site's local MGMT report from LabCorp or MDACC-MDL will then be used to stratify the patient; a post-stratification MGMT central review will be performed, but step 2 registration and protocol treatment can proceed without central review of MGMT
      * Patients whose tissue for central pathology review and official LabCorps or MDACC-MDL MGMT result cannot be received by NRG Oncology Biospecimen Bank on or before 40 calendar days after surgery may NOT enroll on this trial, as central pathology review and stratification will not be complete in time for the patient to start treatment within 49 calendar days following surgery
    * If MGMT has not been assessed locally by LabCorps or MDACC-MDL:

      * Tissue for central pathology review and central MGMT assessment must be received by the NRG Oncology Biospecimen Bank on or before postoperative calendar day 30
      * Central MGMT analysis will be performed at MDACC-MDL and used for patient stratification; results will be conveyed to NRG Oncology within 10 business days of receipt of the tissue
      * Patients who have not had local MGMT assessment by LabCorps or MDACC-MDL and whose tissue for central pathology review cannot be received by NRG Oncology Biospecimen Bank on or before 30 calendar days after surgery may NOT enroll on this trial, as central pathology review and stratification will not be complete in time for the patient to start treatment within 49 calendar days following surgery
  * Tissue Requirements:

    * Patients must have at least 1 block of tumor tissue; submission of 2 blocks is strongly encouraged to maximize the chances of eligibility; in total, at least 1 cubic centimeter of tissue composed primarily of tumor must be present
    * Submission of an accompanying hematoxylin and eosin H&E slide(s) is MANDATORY
    * Diagnosis must be made by surgical excision, either partial or complete; stereotactic biopsy and cavitronic ultrasonic surgical (CUSA) techniques are not allowed
* The tumor must be located in the supratentorial compartment only (any component involving the brain stem or cerebellum is not allowed)
* Patients must provide study-specific informed consent prior to step 1 registration
* PRIOR TO STEP 2 REGISTRATION
* Histologically proven diagnosis of glioblastoma (World Health Organization [WHO] grade IV) confirmed by central review prior to step 2 registration
* Tumor tissue that is determined by central pathology review prior to step 2 registration to be of sufficient quantity for central analysis of MGMT status
* History/physical examination within 28 days prior to step 2 registration
* The patient must have recovered from effects of surgery, postoperative infection, and other complications within 28 days prior to step 2 registration
* Documentation of steroid doses within 28 days prior to step 2 registration
* Karnofsky performance status >= 70 within 28 days prior to step 2 registration
* Age >= 18
* Complete blood count (CBC)/differential obtained within 28 days prior to step 2 registration
* Absolute neutrophil count (ANC) >= 1,500 cells/mm^3 (obtained within 28 days prior to step 2 registration)
* Platelets >= 100,000 cells/mm^3 (obtained within 28 days prior to step 2 registration)
* Hemoglobin >= 10.0 g/dl (obtained within 28 days prior to step 2 registration) (note: the use of transfusion or other intervention to achieve hemoglobin [Hgb] >= 10.0 g/dl is acceptable)
* Bilirubin =< 1.5 upper limit of normal (ULN) (within 28 days prior to step 2 registration)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 3 x ULN (within 28 days prior to step 2 registration)
* Negative serum pregnancy test obtained for females of child-bearing potential within 28 days prior to step 2 registration
* As of Amendment 2, if the registering site is a photon center (registering patients to group I), the patient must agree to participate in the advanced imaging sub-study

Exclusion Criteria:

* Prior invasive malignancy (except non-melanomatous skin cancer) unless disease-free for a minimum of 3 years; (for example, carcinoma in situ of the breast, oral cavity, or cervix are all permissible)
* Recurrent or multifocal malignant gliomas
* Any site of distant disease (for example, drop metastases from the GBM tumor site)
* Prior chemotherapy or radiosensitizers for cancers of the head and neck region; note that prior chemotherapy for a different cancer is allowable (except temozolomide)
* Prior use of Gliadel wafers or any other intratumoral or intracavitary treatment are not permitted
* Prior radiotherapy to the head or neck (except for T1 glottic cancer), resulting in overlap of radiation fields
* Severe, active co-morbidity, defined as follows:

  * Unstable angina at step 2 registration
  * Transmural myocardial infarction within the last 6 months prior to step 2 registration
  * Evidence of recent myocardial infarction or ischemia by the findings of S-T elevations of >= 2 mm using the analysis of an electrocardiogram (EKG) performed within 28 days prior to step 2 registration (Note: EKG to be performed only if clinical suspicion of cardiac issue)
  * New York Heart Association grade II or greater congestive heart failure requiring hospitalization within 12 months prior to step 2 registration
  * Serious and inadequately controlled arrhythmia at step 2 registration
  * Serious or non-healing wound, ulcer or bone fracture or history of abdominal fistula, intra-abdominal abscess requiring major surgical procedure, open biopsy or significant traumatic injury within 28 days prior to step 2 registration, with the exception of the craniotomy for surgical resection
  * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of step 2 registration
  * Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects; note, however, that laboratory tests for coagulation parameters are not required for entry into this protocol
  * Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of step 2 registration
  * Acquired immune deficiency syndrome (AIDS) based upon current Centers for Disease Control and Prevention (CDC) definition; note, however, that human immunodeficiency virus (HIV) testing is not required for entry into this protocol; the need to exclude patients with AIDS from this protocol is because the treatments involved in this protocol may be significantly immunosuppressive with potentially fatal outcomes in patients already immunosuppressed
  * Any other severe immunocompromised condition
  * Active connective tissue disorders, such as lupus or scleroderma, that in the opinion of the treating physician may put the patient at high risk for radiation toxicity
  * End-stage renal disease (ie, on dialysis or dialysis has been recommended)
  * Any other major medical illnesses or psychiatric treatments that in the investigator's opinion will prevent administration or completion of protocol therapy
* Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception; this exclusion is necessary because the treatment involved in this study may be significantly teratogenic
* Patients treated on any other therapeutic clinical protocols within 30 days prior to step 2 registration
* Inability to undergo MRI (e.g., due to safety reasons, such as presence of a pacemaker, or severe claustrophobia)
* Postoperative tumor plus surgical bed size exceeds 5 cm in maximum diameter

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 606 (Estimated)
Dates: Start 2014-12-04 (Actual); Primary Completion 2025-07-07 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | Date of randomization to the date of death due to any cause, assessed up to 5 years
  Will be compared between dose-escalated and -intensified photon intensity-modulated radiation therapy or proton beam therapy with concomitant and adjuvant temozolomide and the standard-dose photon irradiation with concomitant and adjuvant temozolomide. The proportion of patients alive will be estimated using the Kaplan-Meier method.

SECONDARY OUTCOMES:
Overall survival | Date of randomization to the date of death, assessed up to 5 years
  Will be compared between dose-escalated and -intensified photon intensity-modulated radiation therapy to dose-escalated and -intensified proton beam therapy. If the instrumental variable assumptions hold, overall survival rate will be estimated using the Kaplan-Meier method.
Progression-free survival | Date of randomization to the date of progression or death, assessed up to 5 years
  Progression-free survival rates will be estimated using the Kaplan-Meier method.
Incidence of treatment-related toxicity, as measured by the Common Terminology Criteria for Adverse Events version 4 | Up to 5 years
  The number and frequency of observed severities of toxicities (grade 3+) by arm will be reported.
Change in perceived cognitive function, as measured by M.D. Anderson Symptom Inventory Brain Tumor | Baseline to up to 60 weeks
  The mean changes from baseline to each follow-up time point for the perceived cognitive symptom severity score.
Change in neurocognitive function, as measured by Hopkins' Verbal Learning Test-Revised, Trail Making Test Parts A and B, and Controlled Oral Word Association Test | Baseline to up to 60 weeks
  The mean changes from baseline to each follow-up time point for the standardized Hopkins' Verbal Learning Test-Revised, Trail Making Test Parts A and B, Controlled Oral Word Association Test and the Clinical Trial Battery composite score.

OTHER OUTCOMES:
CD4 lymphopenia count | Baseline to up to 5 years
  Mean CD4 lymphopenia count change from baseline to each follow-up collection timepoint.
Use of magnetic resonance diffusion and perfusion imaging to differentiate between tumor progression and pseudo-progression | Baseline - cycle 4
  Will be determined retrospectively following central review by an experienced neuro-radiologist blinded to the patient's outcome.
Use of magnetic resonance diffusion and perfusion imaging as early predictors of overall survival | Baseline up to 12 months
  Cox proportional hazard model will be used to analyze the effect of imaging markers on overall survival. Known prognostic factors and patient baseline characteristics will be included in the multivariate analyses as covariates.

CONTACTS AND LOCATIONS:
Overall Officials: Minesh P Mehta, Principal Investigator — NRG Oncology
Locations (237):
- United States (230):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Saint Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Arizona Oncology Associates-West Orange Grove, Tucson, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - AIS Cancer Center at San Joaquin Community Hospital, Bakersfield, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - Eden Hospital Medical Center, Castro Valley, California
  - Fresno Cancer Center, Fresno, California
  - Marin General Hospital, Greenbrae, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - Memorial Medical Center, Modesto, California
  - Kaiser Permanente Oakland-Broadway, Oakland, California
  - Saint Joseph Hospital - Orange, Orange, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Pomona Valley Hospital Medical Center, Pomona, California
  - Kaiser Permanente-Rancho Cordova Cancer Center, Rancho Cordova, California
  - Rohnert Park Cancer Center, Rohnert Park, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - The Permanente Medical Group-Roseville Radiation Oncology, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - South Sacramento Cancer Center, Sacramento, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Kaiser Permanente Cancer Treatment Center, South San Francisco, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - John Muir Medical Center-Walnut Creek, Walnut Creek, California
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Boca Raton Regional Hospital, Boca Raton, Florida
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - University of Florida Health Science Center - Jacksonville, Jacksonville, Florida
  - Baptist Medical Center South, Jacksonville, Florida
  - Miami Cancer Institute, Miami, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Emory Proton Therapy Center, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Northwestern University, Chicago, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Rush MD Anderson Cancer Center, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Radiation Oncology Associates PC, Fort Wayne, Indiana
  - Parkview Hospital Randallia, Fort Wayne, Indiana
  - Parkview Regional Medical Center, Fort Wayne, Indiana
  - IU Health Methodist Hospital, Indianapolis, Indiana
  - Community Cancer Center East, Indianapolis, Indiana
  - Community Cancer Center South, Indianapolis, Indiana
  - Community Cancer Center North, Indianapolis, Indiana
  - IU Health Ball Memorial Hospital, Muncie, Indiana
  - Mercy Hospital, Cedar Rapids, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Norton Hospital Pavilion and Medical Campus, Louisville, Kentucky
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Willis-Knighton Medical and Cancer Center, Shreveport, Louisiana
  - Maryland Proton Treatment Center, Baltimore, Maryland
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - UM Upper Chesapeake Medical Center, Bel Air, Maryland
  - Central Maryland Radiation Oncology in Howard County, Columbia, Maryland
  - UM Baltimore Washington Medical Center/Tate Cancer Center, Glen Burnie, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Mass General/North Shore Cancer Center, Danvers, Massachusetts
  - Lowell General Hospital, Lowell, Massachusetts
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - McLaren Cancer Institute-Bay City, Bay City, Michigan
  - Corewell Health Dearborn Hospital, Dearborn, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - McLaren Cancer Institute-Flint, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - McLaren Cancer Institute-Lapeer Region, Lapeer, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - McLaren Cancer Institute-Macomb, Mount Clemens, Michigan
  - McLaren Cancer Institute-Central Michigan, Mount Pleasant, Michigan
  - McLaren Cancer Institute-Owosso, Owosso, Michigan
  - McLaren Cancer Institute-Northern Michigan, Petoskey, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Corewell Health Beaumont Troy Hospital, Troy, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Saint Luke's Hospital of Duluth, Duluth, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - North Kansas City Hospital, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Capital Health Medical Center-Hopewell, Pennington, New Jersey
  - ProCure Proton Therapy Center-Somerset, Somerset, New Jersey
  - Virtua Voorhees, Voorhees Township, New Jersey
  - New York-Presbyterian/Brooklyn Methodist Hospital, Brooklyn, New York
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Mission Hospital, Asheville, North Carolina
  - Novant Health Forsyth Medical Center, Winston-Salem, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Cleveland Clinic Akron General, Akron, Ohio
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Geauga Hospital, Chardon, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Mercy Cancer Center-Elyria, Elyria, Ohio
  - Cleveland Clinic Cancer Center Independence, Independence, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - UH Seidman Cancer Center at Southwest General Hospital, Middleburg Heights, Ohio
  - University Hospitals Parma Medical Center, Parma, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - UH Seidman Cancer Center at Firelands Regional Medical Center, Sandusky, Ohio
  - Cleveland Clinic Cancer Center Strongsville, Strongsville, Ohio
  - University of Toledo, Toledo, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - UHHS-Westlake Medical Center, Westlake, Ohio
  - Cleveland Clinic Wooster Family Health and Surgery Center, Wooster, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Willamette Valley Cancer Center, Eugene, Oregon
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Saint Luke's University Hospital-Bethlehem Campus, Bethlehem, Pennsylvania
  - Northeast Radiation Oncology Center, Dunmore, Pennsylvania
  - Ephrata Cancer Center, Ephrata, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - UPMC Pinnacle Cancer Center/Community Osteopathic Campus, Harrisburg, Pennsylvania
  - Sechler Family Cancer Center, Lebanon, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Jefferson Torresdale Hospital, Philadelphia, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - WellSpan Health-York Cancer Center, York, Pennsylvania
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Self Regional Healthcare, Greenwood, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Tennessee Cancer Specialists-Dowell Springs, Knoxville, Tennessee
  - Dell Seton Medical Center at The University of Texas, Austin, Texas
  - Austin Cancer Centers-Central Austin, Austin, Texas
  - Texas Oncology-Austin Midtown, Austin, Texas
  - Texas Oncology - Central Austin Cancer Center, Austin, Texas
  - Texas Oncology - South Austin Cancer Center, Austin, Texas
  - Austin Cancer Centers-North, Austin, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Texas Oncology - Denison Cancer Center, Denison, Texas
  - Texas Oncology-Flower Mound, Flower Mound, Texas
  - Texas Oncology - Fort Worth Cancer Center, Fort Worth, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Memorial Hermann Memorial City Medical Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - UTMB Cancer Center at Victory Lakes, League City, Texas
  - Covenant Medical Center-Lakeside, Lubbock, Texas
  - Texas Oncology-Seton Williamson, Round Rock, Texas
  - Texas Oncology - Round Rock Cancer Center, Round Rock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Texas Oncology Cancer Center Sugar Land, Sugar Land, Texas
  - Texas Oncology - Tyler, Tyler, Texas
  - Logan Regional Hospital, Logan, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Saint George Regional Medical Center, St. George, Utah
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont Medical Center, Burlington, Vermont
  - Dartmouth Cancer Center - North, Saint Johnsbury, Vermont
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - FHCC at Northwest Hospital, Seattle, Washington
  - FHCC Proton Therapy Center, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - Compass Oncology Vancouver, Vancouver, Washington
  - Legacy Salmon Creek Hospital, Vancouver, Washington
  - Wheeling Hospital/Schiffler Cancer Center, Wheeling, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Froedtert Menomonee Falls Hospital, Menomonee Falls, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
- Canada (7):
  - BCCA-Vancouver Island Cancer Centre, Victoria, British Columbia
  - Ottawa Hospital and Cancer Center-General Campus, Ottawa, Ontario
  - Windsor Regional Cancer Centre, Windsor, Ontario
  - CHUM - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - The Research Institute of the McGill University Health Centre (MUHC), Montreal, Quebec
  - CHU de Quebec-L'Hotel-Dieu de Quebec (HDQ), Québec, Quebec
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan